CLINICAL TRIAL: NCT04996121
Title: The Safety Tolerability Pharmacokinetic Characteristics and Efficacy of XZP-5955 Tablets in Patients With NTRK or ROS1 Gene Fusion Locally Advanced or Metastatic Solid Tumors in a Single-arm Open-label Multi-center Phase I/II Clinical Study
Brief Title: A Study of XZP-5955 Tablets in Patients With NTRK or ROS1 Fusion Positive Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZP-5955-1001
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; Locally Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: XZP-5955; Safety, tolerability, pharmacokinetics and efficacy; Solid tumors with NTRK or ROS1 gene fusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XZP-5955 tablets (Experimental): XZP-5955 tablets
  Interventions: Drug: XZP-5955 tablets

INTERVENTIONS:
Drug: XZP-5955 tablets — Phase I dose escalation:
  For each dose cohort, XZP-5955 tablet will be administered orally, single dose for day 1 and then from day 4, administered for continuous cycles of 21 consecutive days for each cycle
  Phase I dose expansion:
  XZP-5955 tablet will be administered orally, once daily for continuous cycles of 21 consecutive days for each cycle. Some patients for PK sample collection, the drug will be administered single dose for day 1, then from day 4, administered for continuous cycles of 21 consecutive days for each cycle
  Phase II:
  XZP-5955 tablet will be administered orally, once daily for continuous cycles of 21 consecutive days for each cycle

SUMMARY:
A phase I/II study to examine the safety, tolerability, pharmacokinetics and efficacy of XZP-5955 tablets in patients with advanced solid tumors harboring NTRK or ROS1 gene fusion

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years old;
2. Phase I dose escalation period: Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic solid tumor, assessed by investigator that no standard therapy exists, or the tumor has relapsed, progressed or was nonresponsive to available therapies, or intolerance, or not suitable to standard therapy at current stage. Priority will be given to patients who have previously documented NTRK or ROS1 gene fusion confirmed by the central laboratory; Phase I dose expansion and Phase II: Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic solid tumor, patients can provide a written report of pathological diagnosis of NTRK or ROS1 positive tested by qualified laboratory;
3. Phase I dose expansion cohort 1 and Phase II cohort 1: locally advanced, or metastatic solid tumor with NTRK gene fusion Phase I dose expansion cohort 2 and Phase II cohort 2： locally advanced, or metastatic NSCLC with ROS1 gene fusion that has progressed to crizotinib and other therapies or was intolerance to crizotinib Phase I dose expansion cohort 3: locally advanced, or metastatic NSCLC with ROS1 gene fusion who have not previously received crizotinib or other therapy.
4. phase I dose escalation: at least 1 measurable target lesion according to RECIST version 1.1 Phase I dose expansion and Phase II: at least 1 measurable target lesion according to RECIST version 1.1 (Tumor lesions treated with prior radiation or other local treatment are considered measurable if they show definite progression)
5. ECOG PS 0-1
6. Life expectancy ≥ 3 months.
7. Adequate organ function:

   Baseline laboratory values fulfilling the following requirements: Absolute neutrophils count (ANC) ≥1.5 × 109/L; Platelets (PLTs) ≥75 × 109/L; Hemoglobin ≥ 85g/L; Serum creatinine≤ 1.5 × ULN， or creatinine clearance ≥50 mL/min/1.73m2(only when serum creatinine>1.5 × ULN); Total serum bilirubin ≤1.5 × ULN; Liver transaminases (AST/ALT) ≤ 2.5 × ULN，≤3× ULN if liver metastases are present or liver cancer patients; Activated Partial Thromboplastin Time≤1.5× ULN；International Normalized Ratio (INR)≤1.5× ULN；
8. Eligible patients (male and female) who are fertile must agree to at least use a reliable contraceptive method with partner during the trial and within 90 days from the last dose; Women of childbearing age must have a negative serum pregnancy test within 7 days before the first dose of the trial.

Exclusion Criteria:

1. Received anti-tumor therapy such as chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy or other therapy within 4 weeks prior to the first dose of the investigational drug except the following:

   Nitroso ureas or mitomycin C within 6 weeks before the first dose of the drug; Oral fluorouracil and small molecule targeted drugs within 2 weeks prior to the first dose of drug or within 5 half life (whichever is longer);
2. Received other unmarketed investigational drugs or treatments within 4 weeks prior to the first dose of the investigational drug;
3. Major organ surgery (except biopsy) or significant trauma within 4 weeks prior to first dose of the investigational drug or required elective surgery during the trial;
4. Adverse reactions to previous antitumor therapy have not recovered to NCI CTCAE 5.0 ≤ grade 1 (except for alopecia, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy, etc.);
5. Inability to swallow drug, or a condition that the investigator judged to severely affect gastrointestinal absorption (eg:Chronic Diarrhea, intestinal obstruction, etc.);
6. Cerebral or meningeal metastases with clinical symptoms. The below patients were allowed to be included: those who were asymptomatic, stable, and did not require steroid treatment for more than 4 weeks prior to the start of study treatment (if the cerebral metastases had undergone radiotherapy or/and surgery, radiotherapy and surgery should be at least 1 month prior to the first dose) ;
7. Known active infections and currently need intravenous anti-infective therapy;
8. History of immune deficiencies, including positive HIV antibody tests;
9. Active Hepatitis B (HBsAg and/or HBcAb positive with HBV-DNA > 500IU/ml) or hepatitis c virus infection (positive test results of anti-HCV with positive HCV-RNA );
10. Known interstitial lung disease (except for radioactive pulmonary fibrosis that does not require steroid therapy);
11. History of serious cardiovascular disease;
12. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I dose escalation) | 24days following first dose of XZP-5955
  Determine MTD of XZP-5955
Number of patients with adverse events (Phase I dose escalation) | within 30 days from last dose
  Incidence of AE as assessed by CTCAE 5.0
Overall Response Rate (ORR) by Blinded Independent Central Review (BICR) (Phase I dose expansion and phase II) | 2 to 3 years after first dose of XZP-5955
  Per RECIST v1.1 as assessed by BICR

SECONDARY OUTCOMES:
Phase I: Area under the concentration versus time curve of XZP-5955 in plasma (AUC) | Pre-dose, up to 72h after drug on Day 1；pre-dose on day 8, day 15 of cycle 1, , pre-dose and up to 12h after drug on day21 of cycle 1;pre-dose on day1 of cycle 2 and 3
  To determine the area under the plasma concentration time curve (AUC) of XZP-5955
Phase I: Maximum plasma concentration (Cmax) of XZP-5955 | Up to 72 hours post dose of Day 1
  To determine the maximum plasma concentration (Cmax) of XZP-5955
Phase I: Oral clearance (CL/F) of XZP-5955 | Pre-dose, up to 72h after drug on Day 1；pre-dose on day 8, day 15 of cycle 1, pre-dose and up to 12h after drug on day21 of cycle 1;pre-dose on day1 of cycle 2 and 3
  To determine the oral clearance (CL/F) of XZP-5955
objective response rate (ORR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the preliminary objective response rate (ORR) by investigator
Progression free survival (PFS) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the PFS by BICR and investigator
Duration of response (DOR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the DOR by BICR and investigator
Disease control rate (DCR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the DOR by BICR and investigator
Clinical benefit rate (CBR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the CBR by BICR and investigator
Time to response (TTR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the TTR by BICR and investigator
Death of response (DpR) (Phase I and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the DpR by BICR and investigator
Overall survival (OS) (Phase I expansion period and Phase II) | 2 to 3 years after first dose of XZP-5955
  To determine the OS
Intracranial objective response rate (Phase I expansion period and Phase II) | To determine the intracranial ORR
  2 to 3 years after first dose of XZP-5955
Number of patients with adverse events ((Phase I dose expansion and Phase II) | within 30 days from last dose
  Incidence of AE as assessed by CTCAE 5.0
Pop PK of XZP-5955 and its metabolite (Phase II) | pre-dose, Tmax on Day1, pre-dose on day 8 of cycle 1, pre-dose on day 1 of Cycle 2, Tmax,ss on Day 1 of cycle 2, pre-dose on day 1 of cycle 3
  To determine the PopPK characteristics of XZP-5955

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China